CLINICAL TRIAL: NCT03347162
Title: Prognostic Role of Muscle Dysfunction in Patients With Gastrointestinal or Hepatobiliary Cancer - An Observational Study of Two Patient Cohorts
Brief Title: Muscle Dysfunction in Gastrointestinal or Hepatobiliary Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jesper Frank Christensen, PhD, Senior researcher, Rigshospitalet, Denmark
Other Study IDs: MuscleLab1.0
Record Dates: First submitted 2017-10-12; First posted 2017-11-20 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Cancer; Cancer of Pancreas; Cancer of Liver; Cancer of Esophagus; Cancer of Stomach; Cancer, Metastatic
Keywords: Cancer; Muscle mass; Muscle strength; Complications; Patient reported outcomes; PRO; Physical function
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be immediately analyzed for plasma biochemistry and a 10 ml plasma sample will be frozen and stored in a study specific biobank.
  As an optional procedure (amendment), we will collect biological tissue from tumor (1mg), muscle (200 mg) and fat (200 mg) biopsies during surgery, from which RNA will be extracted and used to assess small RNA and gene expression by microarray technology and quantitative PCR. For the optional procedure, patients will sign additional separate informed consent before any biopsies are taken. This material will be stored in a study specific biobank until the study is completed, expected 31.12.2022
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 - Resectable patients: These patients will undergo 3 assessments: a baseline-assessment prior to surgery, a post-surgery assessment (2 week post-surgery) and a follow-up assessment 6 months after surgery (after adjuvant oncology treatment).
- Cohort 2 - Non-resectable patients: These patients will undergoing 3 assessments: a baseline-assessment prior to palliative treatment, an acute measurement 4 weeks after initiation of palliative treatment, and a 6-month long-term assessment.

SUMMARY:
PURPOSE: To determine the prognostic properties of a comprehensive evaluation of body composition and physical function in patients with GI-HEP cancer from point of diagnosis and throughout the treatment trajectory.

GI-HEP: Patients with tumors of the upper gastrointestinal or hepatobiliary tract, specifically tumors of the esophagus, gastro-esophageal junction, stomach, primary tumors of the liver or biliary tract, as well as colorectal liver metastasis or tumors of the pancreas.

DETAILED DESCRIPTION:
RATIONAL: Patients diagnosed with GI-HEP cancer are faced with poor prognosis. The treatment is demanding and associated with severe deconditioning potentially leading to worse prognostic outcomes. To what extend patients body composition at the point of diagnoses, as well as changes in body composition throughout the cancer continuum is associated with cancer outcomes is currently not well-described, specifically if this should be part of standard clinical evaluation in order to optimize therapy-efficacy. Recent findings suggest that pathophysiological alterations in skeletal muscle mass and function can have significant implications for the risk of disease progression and long-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with histologically verified GI-HEP cancer

Exclusion Criteria:

* Age: <18
* Pregnancy
* Physical or mental disabilities precluding physical testing
* Inability to read and understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GI-HEP cancer specified as tumors of the esophagus, gastroesophageal junction, stomach, primary tumors of the liver and biliary tract. As well as colorectal liver metastasis and tumors of the pancreas.
  The study will include patients who are candidates for tumor resection and patients who are not candidates for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Post-operative complications | From baseline to 30 days post surgery
  Incidens rate of post-operative complications (Clavien-Dindo grade 2 or higher).
Cohort 2: Medical treatment complications | From baseline to 1 year follow-up
  Incidens rate of medical complications (dose-reduction, temporary or permanent discontinuation)

SECONDARY OUTCOMES:
Hospitalization duration | From baseline to 1 year follow-up
  Total number days in hospital
Disease free survival | From baseline to 1 year follow-up
  Risk of disease progression
Overall survival | From baseline to 1 year follow-up
  Risk of mortality from any-cause
Change in whole body lean mass | From baseline to 6 months follow-up
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in appendicular lean mass | From baseline to 6 months follow-up
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in whole body fat percentage | From baseline to 6 months follow-up
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in visceral fat mass | From baseline to 6 months follow-up
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in bone mineral density | From baseline to 6 months follow-up
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in bone mineral content | From baseline to 6 months follow-up
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in Skeletal Muscle Index | From baseline to 6 months follow-up
  L3 muscle area determined by Computed tomography scan (performed for clinical purpose) adjusted for hight
Change in Walking capacity | From baseline to 6 months follow-up
  Maximum 10 meter walking speed
Change in stair-climbing capacity | From baseline to 6 months follow-up
  Timed Stair-climbing test
Change in lower body physical function | From baseline to 6 months follow-up
  30 seconds Sit-To-Stand test
Change in maximum leg power | From baseline to 6 months follow-up
  Leg extensor power test (Nottingham Power rig)
Change in hand grip strength | From baseline to 6 months follow-up
  Maximum strength test by handgrip dynanometer
Change in plasma total cholesterol concentration | From baseline to 6 months follow-up
  Blood sample
Change in plasma HDL cholesterol | From baseline to 6 months follow-up
  Blood sample
Change in plasma LDL cholesterol | From baseline to 6 months follow-up
  Blood sample
Change in plasma triglycerides | From baseline to 6 months follow-up
  Blood sample
Change in plasma HbA1C | From baseline to 6 months follow-up
  Blood sample
Change in plasma glucose | From baseline to 6 months follow-up
  Blood sample
Change in plasma insulin | From baseline to 6 months follow-up
  Blood sample
Change in health-related quality of life | From baseline to 6 months follow-up
  Functional Assessment of Cancer Therapy (FACT) questionnaire
Change in psychological distress | From baseline to 6 months follow-up
  Hospital Anxiety and Depression Scale (HADS) questionnaire
Change in sleep quality | From baseline to 6 months follow-up
  Pittsburgh Sleep Quality Index (PSQI) questionnaire
Change in physical activity level | From baseline to 6 months follow-up
  International Physical Activity Questionnaire (IPAQ) short form

CONTACTS AND LOCATIONS:
Overall Officials: Jesper F Christensen, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark